CLINICAL TRIAL: NCT02972619
Title: Management of Hypertension and Multiple Risk Factors to Enhance Cardiovascular Health - A Cluster Randomized Trial in Singapore Polyclinics
Brief Title: Management of Hypertension and Multiple Risk Factors to Enhance Cardiovascular Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: SingHealth Polyclinics (Other)
Responsible Party: Principal Investigator, Professor Tazeen Jafar, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NMRC/CSA-SI/0005/2015
Record Dates: First submitted 2016-11-20; First posted 2016-11-23 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Hypertension; Cardiovascular Disease
Keywords: Blood Pressure; Lipids; Cardiovascular; Health Services; Hypertension
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Structured multicomponent intervention (MCI)
  Interventions: Other: Structured Multicomponent Intervention (MCI)
- Usual Care (No Intervention): Control group receive usual care in the polyclinics

INTERVENTIONS:
Other: Structured Multicomponent Intervention (MCI) — Multicomponent Intervention (MCI) includes 1) algorithm-driven antihypertensive treatment for all hypertensive individuals using fixed-dose combination (FDC) and lipid lowering for high risk hypertensive individuals, 2) motivational conversation for high-risk hypertensive individuals and 3) telephone based follow-ups of all hypertensive individuals by a team of physician supervised nurse, and 4) discounts on FDC antihypertensive medications
  Arms: Intervention

SUMMARY:
Background: Hypertension is a serious public health problem responsible for significant mortality and morbidity from cardiovascular disease. In Singapore, 1 in 4 adults age 30 years or older suffer from hypertension. Nearly half of these patients have uncontrolled hypertension and only 50% of individuals are on antihypertensive treatment. Our study aims to evaluate the effectiveness, cost effectiveness and impact on medication adherence of a well-structured program using multicomponent intervention for hypertension control aimed at overall cardiovascular risk reduction among individuals with hypertension attending the polyclinics in Singapore, compared to existing services. Such a program is expected to be cost-effective in terms of improving hypertensive individuals' outcomes, and to be potentially scalable and sustainable.

Methods/design: Cluster randomized trial of 8 of the nine SingHealth Polyclinics randomized to intervention or usual care (4 each) and followed up for 2 years post randomization

Intervention: The structured multicomponent primary care program comprises of: 1) algorithm-driven antihypertensive treatment for all hypertensive individuals and using fixed-dose combination (FDC) and lipid-lowering medication for high-risk hypertensive individuals, 2) motivational conversation for high-risk hypertensive individuals, 3) Follow-up of all hypertensive individuals on improving blood pressure (BP) as a primary outcome and other cardiovascular risk factors as a secondary outcome, and 4) discounts on FDC antihypertensive medication

Usual care: The participants attending polyclinics randomized to usual care will continue to receive treatment from the health providers according to existing practices. The hypertensive individuals will also continue to pay for the services (physician or nurse consultation) as per their existing model of reimbursement.

Participants: A total of 1000 participants will be recruited, 125 from each of the 8 polyclinics. Recruitment will be in batches of 4 and 4 clinics sequentially (balanced by randomization group).

Outcomes: All hypertensive individuals will be assessed by trained outcomes assessors independent to treatment at baseline, 1-year and 2-yeat post randomization. The primary outcome will be the change in systolic blood pressure from baseline to 2 years. Primary Cost-Effectiveness measures will be- 1) Incremental cost per mm Hg systolic BP reduction from baseline to end of follow-up at two years post randomization; 2) incremental cost per projected CVD disability adjusted life years (DALYs) averted and quality adjusted life years (QALYs) saved, and 3) incremental cost per change in cardiovascular risk score from baseline to final follow-up at two-year post. The impact of effect on adherence to antihypertensive and lipid medication will be measured using data on adherence obtained from polyclinic pharmacy records and clinic notes. An average of percent adherence to antihypertensive and lipid lowering will be computed as a composite score. The change in percent composite adherence to antihypertensive and lipid medications from baseline to follow up will be compared between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* 40 years or older
* Singapore citizens or Permanent Residents
* Visiting the recruiting polyclinic at least twice during the last 1 year
* Individuals with a diagnosis of hypertension (systolic BP ≥ 140 mm Hg or diastolic BP ≥ 90 mm Hg on two or more prior visits; physician diagnosed hypertension, or on antihypertensive medications) and uncontrolled blood pressure (systolic BP ≥ 140 mm Hg or diastolic BP ≥ 90 mm Hg)

Exclusion Criteria:

* Active systemic illness including fever, recent hospitalization (i.e. during last 4 months),
* Clinically unstable heart failure or advanced kidney disease {estimated CKD-Epi glomerular filtration rate (GFR) <40 ml/min/1.73m2 or nephrotic range proteinuria (i.e. 3g/d or more)},
* Known liver disease,
* Pregnancy or breastfeeding
* Any other major debilitating disease or mental illness that precludes validity of informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-15 (Actual); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure from baseline to final follow-up at 24 months | Baseline to 2 years

SECONDARY OUTCOMES:
Change in serum LDL from baseline to final follow-up at 24 months | Baseline to 2 years
Proportion of hypertensive individuals with BP controlled to target or > 5 mm Hg decrease in systolic BP | Baseline to 2 years
Proportion of hypertensive individuals with decrease in LDL cholesterol by >0.4 mmol/L (>15 mg/dl). | Baseline to 2 years
Composite outcome of death or hospital admission due to Coronary heart disease (CHD), heart failure, or stroke | 2years
Individual outcomes of all-cause mortality, Cardiovascular disease (CVD) deaths, and hospital admission due to CHD, heart failure, or stroke | 2 years
Decrease of > 0.5 percent in glycated hemoglobin or change in proportion of hypertensive individuals with glycated hemoglobin <7% in hypertensive individuals with diabetes | Baseline to 2 years
Change in albuminuria from baseline to follow-up at 24 months | Baseline to 2 years
Change in estimated CKD-EPI GFR from baseline to follow-up at 24 months | Baseline - 2 years
Change in cardiovascular disease (CVD) risk score | Baseline - 2 years
Individual outcomes of change in a) diastolic BP and b) total cholesterol from baseline to end of follow-up at 24 months | Baseline to follow-up 2 years
Change in lifestyle (diet, physical activity based on self-report) or BMI between groups | Baseline to 2 years
Change in systolic blood pressure from baseline to 12 months | Baseline to 1 year
Change in serum LDL cholesterol from baseline to 12 months | Baseline to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tazeen Jafar, MD, MPH, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- SingHealth Polyclinics (SHP), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chay J, Jafar TH, Su RJ, Shirore RM, Tan NC, Finkelstein EA. Cost-Effectiveness of a Multicomponent Primary Care Intervention for Hypertension. J Am Heart Assoc. 2024 Apr 16;13(8):e033631. doi: 10.1161/JAHA.123.033631. Epub 2024 Apr 12. PMID 38606776
- [Derived] Jafar TH, Tan NC, Shirore RM, Allen JC, Finkelstein EA, Hwang SW, Koong AYL, Moey PKS, Kang GC, Goh CWT, Subramanian RC, Thiagarajah AG, Ramakrishnan C, Lim CW, Liu J; for SingHypertension Study Group. Integration of a multicomponent intervention for hypertension into primary healthcare services in Singapore-A cluster randomized controlled trial. PLoS Med. 2022 Jun 13;19(6):e1004026. doi: 10.1371/journal.pmed.1004026. eCollection 2022 Jun. PMID 35696440
- [Derived] Porhcisaliyan VD, Wang Y, Tan NC, Jafar TH. Socioeconomic status and ethnic variation associated with type 2 diabetes mellitus in patients with uncontrolled hypertension in Singapore. BMJ Open Diabetes Res Care. 2021 Jul;9(1):e002064. doi: 10.1136/bmjdrc-2020-002064. PMID 34301679
- [Derived] Allen JC Jr, Halaand B, Shirore RM, Jafar TH; for SingHypertension Study Group. Statistical analysis plan for management of hypertension and multiple risk factors to enhance cardiovascular health in Singapore: the SingHypertension pragmatic cluster randomized controlled trial. Trials. 2021 Jan 19;22(1):66. doi: 10.1186/s13063-020-05016-4. PMID 33468225
- [Derived] Jafar TH, Tan NC, Allen JC, Finkelstein EA, Goh P, Moey P, Quah JHM, Hwang SW, Bahadin J, Thiagarajah AG, Chan J, Kang G, Koong A. Management of hypertension and multiple risk factors to enhance cardiovascular health in Singapore: The SingHypertension cluster randomized trial. Trials. 2018 Mar 14;19(1):180. doi: 10.1186/s13063-018-2559-x. PMID 29540213